CLINICAL TRIAL: NCT07110103
Title: Golidocitinib With PD-1 Inhibitors as Maintenance Treatment in Patients With Previously Untreated Extensive-stage Small Cell Lung Cancer: an Open-label, Single-arm, Phase 2 Study
Brief Title: Golidocitinib With PD-1 Inhibitors as Maintenance Treatment for Previously Untreated ES-SCLC
Acronym: JACKPOT38
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Dizal (Jiangsu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5342
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: SCLC; SCLC, Extensive Stage
Keywords: golidocitinib; ES-SCLC
MeSH Terms: interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- golidocitinib with PD-1 inhibitors (Experimental): Patients will firstly receive 4 cycles of PD-1 inhibitors and chemotherapy as induction treatment, and patients who don't progress during induction period will continue to receive golidocitinib with PD-1 inhibitors as maintenance treatment until disease progression.
  Interventions: Drug: golidocitinib with PD-1 inhibitors

INTERVENTIONS:
Drug: golidocitinib with PD-1 inhibitors — Dose escalation: 75/150mg golidocitinib with PD-1 inhibitors as maintenance treatment after 4 cycles of PD-1 inhibitors and chemotherapy.
  Dose expansion: Selected dose (75mg or 150mg) of golidocitinib with PD-1 inhibitors as maintenance treatment after 4 cycles of PD-1 inhibitors and chemotherapy.
  Other Names: AZD4205

SUMMARY:
This is an open-label, single-arm, phase 2 study to evaluate the safety and efficacy of golidocitinib with PD-1 inhibitors as maintenance treatment in patients with previously untreated extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
This study is a single-arm clinical study to evaluate the safety and efficacy of golidocitinib combined with PD-1 inhibitors in ES-SCLC. The study consists of two parts:

Part A (dose escalation), which will include previously untreated ES-SCLC subjects, aims to explore the safety and tolerability of golidocitinib combined with PD-1 inhibitors in this population and determine the recommended dose of the combination.

Part B (dose expansion), which will include previously untreated ES-SCLC subjects, aims to explore the preliminary efficacy of golidocitinib combined with PD-1 inhibitors in this population and evaluate the efficacy and safety.

After completing the required assessments during the screening period and meeting the eligibility criteria, the subjects will first receive 4 cycles of PD-1 inhibitor combined with chemotherapy in the induction phase, followed by maintenance treatment with PD-1 inhibitor combined with golidocitinib. Subjects will continue to receive PD-1 inhibitor combined with golidocitinib until disease progression, intolerable toxicity, death, withdrawal of informed consent by the subject, or 24 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide a signed and dated informed consent form, including compliance with the requirements and restrictions listed in the ICF and this protocol;
2. Subjects are ≥ 18 years old when signing the ICF;
3. Subjects have an ECOG performance status score of 0 or 1 and have not deteriorated in the past 2 weeks;
4. Life expectancy ≥ 3 months;
5. Histologically or cytologically confirmed ES-SCLC (stage IV [any T stage, any N stage, M1 a/b/c stage] according to the 8th edition of the AJCC TNM staging system for lung cancer, or T3-4 stage disease caused by multiple lung nodules and the disease is too diffuse, or the tumor/nodule volume is too large to be tolerated by a tolerable radiotherapy plan);
6. The presence of at least one measurable lesion (based on RECIST 1.1): with a long diameter ≥ 10 mm (lymph node lesions require a short diameter of ≥15 mm) that can be accurately and repeatedly measured at baseline under CT or MRI; and there are measurable lesions outside the central nervous system;
7. SCLC patients who have not received any systemic anti-tumor treatment for advanced disease; if the patient has received neoadjuvant/adjuvant therapy in the past, the interval between the diagnosis of ES-SCLC and the completion of the last treatment must be at least 6 months;
8. Patients must be suitable for platinum (cisplatin or carboplatin)-based chemotherapy as the first-line treatment for ES-SCLC;
9. Adequate bone marrow reserve and organ system function reserve, summarized as follows:

   * Absolute neutrophil count (ANC) ≥ 1.5×109/L without growth factor support;
   * Platelet ≥ 100×109/L without growth factor support or blood transfusion;
   * Hemoglobin ≥ 9 g/dL or 90 g/L without erythropoietin or blood transfusion;
   * Total bilirubin ≤ 1.5 × ULN; if suffering from Gilbert syndrome (unconjugated hyperbilirubinemia), total bilirubin should be ≤ 3 × ULN;
   * ALT and AST ≤ 2.5 × ULN. For patients with documented liver metastases, AST and ALT levels ≤ 5 × ULN;
   * Creatinine clearance calculated by the Cockcroft-Gault method, >60 ml/min for patients receiving cisplatin and >45 ml/min for patients receiving carboplatin;
   * Urine routine examination shows less than 2+ protein in urine, or 24-hour urine protein quantitative <1 g;
   * Good coagulation function, defined as international normalized ratio (INR) and/or prothrombin time (PT) ≤1.5 times ULN and/or activated partial thromboplastin time (APTT) ≤1.5 upper limit of normal; if the subject is receiving anticoagulant therapy, as long as the PT is within the intended use range of the anticoagulant drug;
   * Serum amylase ≤1.5 times ULN and/or serum lipase ≤1.5 times ULN;
   * Left ventricular ejection fraction (LVEF) ≥ 55%;
10. For patients with central nervous system metastases, the following conditions must be met before they can be included:

    * No neurological symptoms or symptoms are stable for at least 2 weeks after local treatment, no need to use corticosteroids or anti-epileptic drugs, and hormonal treatment has been stopped within 3 days before the first dose of study drug;
    * If brain metastases have been treated locally (radiotherapy or surgery), there should be a time window of ≥ 2 weeks before the first dose of study treatment to ensure that local treatment-related adverse events have been reduced to CTCAE ≤ 1 grade;
11. Women of childbearing potential must undergo a urine and/or serum pregnancy test (if the urine test cannot be confirmed as negative) within 7 days before the first medication, and the result must be negative; WOCBP or men and their WOCBP partners should agree to take effective contraceptive measures from the signing of the ICF until 6 months after the last dose of the study drug;
12. The subjects should be able to understand the study protocol and voluntarily comply with the study and follow-up;
13. For patients who are about to enter the maintenance period, the investigator shall determine whether they are suitable for starting treatment with golidocitinib combined with PD-1 inhibitors (generally all previous toxicities must be alleviated to CTCAE ≤ 1 level, excluding hair loss, fatigue or other conditions that are judged by the investigator to be clinically insignificant).

Exclusion Criteria:

1. Histopathological confirmation of the presence of mixed NSCLC and SCLC components;
2. The presence of spinal cord compression or meningeal metastasis;
3. Any of the following medical histories:

   * Systemic treatment with Chinese patent medicines with anti-lung cancer indications or immunomodulatory drugs (including thymosin, interferon, interleukin, excluding local use for the control of pleural effusion) within 2 weeks before the first dose;
   * Currently participating in interventional clinical research treatment, or receiving other research drugs or using research devices within 4 weeks before the first dose; any drug still in the development stage needs to be washed out for 5 half-lives (or discussed with the research team);
   * Other major surgeries other than diagnosis or biopsy (excluding vascular access) within 4 weeks before the first dose, or major surgery is expected during the study;
   * Palliative radiotherapy within 2 weeks before the first dose;
   * Serious arterial/venous thrombotic events, including cerebrovascular accident (e.g., history of stroke or intracranial hemorrhage), deep vein thrombosis, and pulmonary embolism, occurred within 6 months before the first dose;
   * Currently receiving (or unable to stop taking at least 1 week before the first dose) drugs, herbal supplements, and foods that are known to be strong inducers or inhibitors of CYP3A;
   * Prior to the first dose, there was a CTCAE caused by previous treatment > Grade 1 adverse events (except alopecia of any degree);
4. Receiving solid organ or blood system transplantation (such as previous allogeneic bone marrow transplantation or whole blood transfusion within 120 days of sample collection during the study);
5. Previous interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid hormone treatment, or current clinically active interstitial lung disease (including interstitial lung changes), immune pneumonitis caused by immunotherapy;
6. Active autoimmune disease requiring systemic treatment (such as the use of disease-modifying drugs, corticosteroids or immunosuppressants) within 2 years before the first dose. Replacement therapy (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is not considered systemic treatment;
7. Diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of the study. Physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are allowed;
8. Diagnosed with other malignancies within 5 years before the first dose, excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has been evaluated to be clinically cured;
9. Vaccinated with live vaccines within 30 days before the first dose (cycle 1, day 1), including live attenuated vaccines, excluding inactivated vaccines;
10. Known active tuberculosis, such as positive tuberculin (PPD) test (nodule diameter > 10 mm), positive T-SPOT test, chest X-ray/CT Tuberculosis lesions are found, or other positive results are found based on routine clinical screening (except for those who have been cured after standardized anti-tuberculosis treatment as assessed by the researchers);
11. Subjects currently have severe infectious diseases that are difficult to control and must be excluded. After the recent infectious diseases are under control, the research team must determine whether they can be included in the group;
12. Subjects with active infections, including but not limited to hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) and COVID-19 active infections (determined by the researchers to be clinically significant, with signs or symptoms, etc.). Testing for COVID-19 will be based on local practice;
13. Meet any of the following cardiac criteria:

    * Congestive heart failure (CHF) classified as class II by the New York Heart Association (NYHA);
    * Clinically significant valvular heart disease, hypertrophic or constrictive cardiomyopathy;
    * Any clinically significant abnormalities on resting ECG, such as complete left bundle branch block, 2/3 degree atrioventricular block, PR interval > 250 msec;
    * Average calibrated QTcF > 470 msec of 3 resting ECGs during the screening period;
    * Subjects with any factors that may cause QT prolongation or increased risk of arrhythmic events (e.g., heart failure, hypokalemia, congenital long QT syndrome or a first-degree relative with long QT syndrome or a family history of unexplained sudden death under the age of 40, or any concomitant medication known to cause QT prolongation);
    * Ventricular arrhythmias requiring treatment;
    * Acute myocardial infarction (AMI), unstable angina or new angina within 6 months before the administration of this study;
14. Allergy to the drugs used in the study or their ingredients;
15. Intractable nausea and vomiting, chronic gastrointestinal diseases, difficulty swallowing drugs, intestinal obstruction or previous intestinal resection, which may lead to inability to fully absorb the study drugs;
16. Pregnant or lactating women;
17. Known bleeding diathesis, that is, hemophilia, von Willebrand disease;
18. The investigators assess that there are severe or uncontrollable systemic diseases (including poorly controlled hypertension and bleeding diseases) that cannot be carried out in clinical studies or may lead to poor compliance with clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to the end of monitoring at 2 years
  Time from the subject started treatment to disease progression or death due to any cause based on the investigators' evaluation

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment to the end of monitoring at 2 years
  Time from the subject started treatment to death due to any cause based on the investigators' evaluation
Safety and Tolerability | From enrollment to the end of monitoring at 2 years
  Incidence, nature, and severity of adverse events (AEs), graded according to NCI-CTCAE v5.0, including immune-related AEs and serious AEs

CONTACTS AND LOCATIONS:
Overall Officials: Zhijie Wang, MD, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Xinqiao Hospital, Third Military Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: No